CLINICAL TRIAL: NCT04313972
Title: IC PaIN Trial: Interstitial Cystitis Pain Improvement With Naltrexone, the Effect of Low Dose Naltrexone on Symptoms and Pain of Patients With Interstitial Cystitis/Painful Bladder Syndrome a Randomized Placebo-controlled Prospective Trial
Brief Title: IC PaIN Trial: Interstitial Cystitis Pain Improvement With Naltrexone
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: There was a delay in recruitment initiation due to COVID-19 and internal logistical challenges. Following this delay, the principal investigator left the study site, and it was determined that the study should be terminated.
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Ghazaleh Rostami Nia, Principal Investigator, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EH20-127
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Interstitial Cystitis; Painful Bladder Syndrome; Bladder Pain Syndrome; Low Dose Naltrexone; Low-dose Naltrexone; Naltrexone
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-dose naltrexone (Experimental): 2mg low-dose naltrexone capsules
  Interventions: Drug: low-dose naltrexone
- Placebo (Placebo Comparator): Placebo capsules
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: low-dose naltrexone — 2mg of low-dose naltrexone nightly for 2 weeks, then 4mg of low-dose naltrexone nightly for 4 weeks
  Arms: Low-dose naltrexone
Drug: Placebo oral tablet — 1 capsule nighty for 2 weeks, then 2 capsules nightly for 4 weeks
  Arms: Placebo

SUMMARY:
Interstitial cystitis/painful bladder syndrome (IC/PBS) is a debilitating condition with symptoms of urinary urgency, frequency, nocturia (waking up at night to void), and pain, without evidence of urinary tract infection or other identifiable causes. IC/PBS often coexists with other chronic pain syndromes, such as irritable bowel syndrome, chronic fatigue syndrome, and fibromyalgia.

Several treatments exist for IC/PBS; some are not effective, others are time consuming for patients to receive, some can take weeks to months before they become effective, and many have risks associated with them. Low-dose naltrexone (LDN) has demonstrated improvement of symptoms in conditions associated with IC/PBS. LDN is defined as less than 5mg of naltrexone. Some adverse effects have been reported with LDN, the most common are vivid dreams, nightmares, and insomnia.

The investigators hypothesis LDN will have greater than 30% reduction in symptoms as defined by the Interstitial Cystitis Symptom Index in patients diagnosed with IC/PBS from baseline when compared to placebo. The 30% reduction in pain is a standard outcome measure in the pain literature. This improvement has been seen in prior studies where LDN was used to treat pain syndromes.

This will be a randomized double-blinded placebo-controlled prospective trial. Patients meeting diagnostic criteria for IC/PBS by American Urologic Association (AUA) guidelines will be eligible, and then must then meet all applicable inclusion and exclusion criteria. Study participants will sign a consent, complete several questionnaires, give a blood sample to measure liver function tests, and once at home, complete a 24-hour bladder diary.

Participants will be randomized to receive either placebo or study medication. Participants will be instructed to take one capsule nightly for two weeks, then increase to two capsules nightly for four weeks. They will be given a log to record the date and time they take the medication. All study participants will also receive first-line behavioral therapy for IC/PBS of a bladder diet and bladder drills.

After six weeks, participants will complete a second bladder diary. They will then complete the exit study questionnaires, have a second liver function test, return any unused medication, and meet with their doctor to discuss conventional treatment options for IC/PBS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged eighteen and older
2. Meet criteria for IC/PBS as defined by the American Urology Association as "an unpleasant sensation (pain, pressure, discomfort) perceived to be related to the urinary bladder, associated with lower urinary tract symptoms or more than six weeks duration, in the absence of infection or other identifiable causes" (8)
3. Newly diagnosed and treatment naïve for IC/PBS or previously diagnosed with IC/PBS, but who have no received treatment in the past four weeks. Patient who use anti-inflammatory medication on an as needed basis in the four weeks prior to the study will be included.
4. Have had a cystoscopy in the last 6 months prior to study entry to rule out confounding conditions
5. English speaking
6. Working telephone number
7. Able to provide a blood sample to evaluate liver enzymes
8. Able to attend research visits

Exclusion Criteria:

1. Patients under the age of 18
2. Patients with known liver disease, including total bilirubin >1.2, AST (aspartate aminotransferase) > 32, ALT (alanine transaminase) > 54
3. Patients with known kidney disease
4. Patients who have thyroid disease and who are taking thyroid replacement medications
5. Patients with known neurologic disease affecting bladder function
6. Patients with known bladder or urethral cancer
7. Patients with bladder, urethral, or ureteral calculi
8. Patients who have had a positive urine culture or a clinical UTI (Urinary Tract Infection) in the past 6 weeks
9. Patients who are currently pregnant or breast feeding (15)
10. Patients who are actively using opioid analgesics
11. Patients with moderate-severe alcohol use disorder
12. Patients who are actively using sleep aids
13. Patients who are regularly using anti-inflammatory medications, such as daily Celebrex for arthritis. Those who use an anti-inflammatory medication on an as needed basis may use the medication prior to enrollment in the study.
14. Patients who have had a known adverse reaction to naltrexone
15. Patients who are acutely ill
16. Patients who are diagnosed with a significant psychological comorbidity that would interfere with study participation (32)
17. Patients who have had a bladder instillation or had oral medical treatment for IC/PBS in the past four weeks.
18. Patients diagnosed with other chronic pelvic pain syndromes, such as endometriosis
19. Patients who are unable to swallow pills/capsules
20. Patients who have had previous treatment with low-dose naltrexone
21. Patients who have previously scheduled surgeries or procedure during the study time period that would require analgesia.
22. Patients who are sexually active and of childbearing potential who are unwilling to use an established and reliable form of contraception for the duration of the study.
23. Patients who are unwilling to have a serum blood test to assess serum transaminases and serum bilirubin.

Ages: 18 Years to 110 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-02-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Pelvic Health at the NorthShore University HealthSystem, Skokie, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Konkle KS, Berry SH, Elliott MN, Hilton L, Suttorp MJ, Clauw DJ, Clemens JQ. Comparison of an interstitial cystitis/bladder pain syndrome clinical cohort with symptomatic community women from the RAND Interstitial Cystitis Epidemiology study. J Urol. 2012 Feb;187(2):508-12. doi: 10.1016/j.juro.2011.10.040. Epub 2011 Dec 15. PMID 22177158
- [Background] Hanno PM, Burks DA, Clemens JQ, Dmochowski RR, Erickson D, Fitzgerald MP, Forrest JB, Gordon B, Gray M, Mayer RD, Newman D, Nyberg L Jr, Payne CK, Wesselmann U, Faraday MM; Interstitial Cystitis Guidelines Panel of the American Urological Association Education and Research, Inc. AUA guideline for the diagnosis and treatment of interstitial cystitis/bladder pain syndrome. J Urol. 2011 Jun;185(6):2162-70. doi: 10.1016/j.juro.2011.03.064. Epub 2011 Apr 16. PMID 21497847
- [Background] Clauw DJ, Schmidt M, Radulovic D, Singer A, Katz P, Bresette J. The relationship between fibromyalgia and interstitial cystitis. J Psychiatr Res. 1997 Jan-Feb;31(1):125-31. doi: 10.1016/s0022-3956(96)00051-9. PMID 9201654
- [Background] Tripp DA, Nickel JC, Wong J, Pontari M, Moldwin R, Mayer R, Carr LK, Doggweiler R, Yang CC, Mishra N, Nordling J. Mapping of pain phenotypes in female patients with bladder pain syndrome/interstitial cystitis and controls. Eur Urol. 2012 Dec;62(6):1188-94. doi: 10.1016/j.eururo.2012.05.023. Epub 2012 May 18. PMID 22633363
- [Background] Nickel JC, Tripp DA, Pontari M, Moldwin R, Mayer R, Carr LK, Doggweiler R, Yang CC, Mishra N, Nordling J. Interstitial cystitis/painful bladder syndrome and associated medical conditions with an emphasis on irritable bowel syndrome, fibromyalgia and chronic fatigue syndrome. J Urol. 2010 Oct;184(4):1358-63. doi: 10.1016/j.juro.2010.06.005. Epub 2010 Aug 17. PMID 20719340
- [Background] Peters K, Diokno A, Steinert B, Yuhico M, Mitchell B, Krohta S, Gillette B, Gonzalez J. The efficacy of intravesical Tice strain bacillus Calmette-Guerin in the treatment of interstitial cystitis: a double-blind, prospective, placebo controlled trial. J Urol. 1997 Jun;157(6):2090-4. PMID 9146587
- [Background] Propert KJ, Payne C, Kusek JW, Nyberg LM. Pitfalls in the design of clinical trials for interstitial cystitis. Urology. 2002 Nov;60(5):742-8. doi: 10.1016/s0090-4295(02)01775-2. No abstract available. PMID 12429288
- [Background] Oh-Oka H. Clinical Efficacy of 1-Year Intensive Systematic Dietary Manipulation as Complementary and Alternative Medicine Therapies on Female Patients With Interstitial Cystitis/Bladder Pain Syndrome. Urology. 2017 Aug;106:50-54. doi: 10.1016/j.urology.2017.02.053. Epub 2017 Apr 20. PMID 28435032
- [Background] O'Leary MP, Sant GR, Fowler FJ Jr, Whitmore KE, Spolarich-Kroll J. The interstitial cystitis symptom index and problem index. Urology. 1997 May;49(5A Suppl):58-63. doi: 10.1016/s0090-4295(99)80333-1. PMID 9146003
- [Background] Korting GE, Smith SD, Wheeler MA, Weiss RM, Foster HE Jr. A randomized double-blind trial of oral L-arginine for treatment of interstitial cystitis. J Urol. 1999 Feb;161(2):558-65. PMID 9915448
- [Background] Parsons CL, Benson G, Childs SJ, Hanno P, Sant GR, Webster G. A quantitatively controlled method to study prospectively interstitial cystitis and demonstrate the efficacy of pentosanpolysulfate. J Urol. 1993 Sep;150(3):845-8. doi: 10.1016/s0022-5347(17)35629-x. PMID 7688432
- [Background] Hanno PM, Wein AJ, Kavoussi LR, Partin AW, Peters C, eds. Bladder pain syndrome (interstitial cystitis) and related disorder. 11th ed. Campbell-Walsh urology. Inc Philadelphia, PA: Elsevier; 2016: 334-370.
- [Background] Anderson VR, Perry CM. Pentosan polysulfate: a review of its use in the relief of bladder pain or discomfort in interstitial cystitis. Drugs. 2006;66(6):821-35. doi: 10.2165/00003495-200666060-00006. PMID 16706553
- [Background] Foster HE Jr, Hanno PM, Nickel JC, Payne CK, Mayer RD, Burks DA, Yang CC, Chai TC, Kreder KJ, Peters KM, Lukacz ES, FitzGerald MP, Cen L, Landis JR, Propert KJ, Yang W, Kusek JW, Nyberg LM; Interstitial Cystitis Collaborative Research Network. Effect of amitriptyline on symptoms in treatment naive patients with interstitial cystitis/painful bladder syndrome. J Urol. 2010 May;183(5):1853-8. doi: 10.1016/j.juro.2009.12.106. Epub 2010 Mar 29. PMID 20303115
- [Background] Parsons CL, Greenberger M, Gabal L, Bidair M, Barme G. The role of urinary potassium in the pathogenesis and diagnosis of interstitial cystitis. J Urol. 1998 Jun;159(6):1862-6; discussion 1866-7. doi: 10.1016/S0022-5347(01)63178-1. PMID 9598476
- [Background] van Ophoven A, Pokupic S, Heinecke A, Hertle L. A prospective, randomized, placebo controlled, double-blind study of amitriptyline for the treatment of interstitial cystitis. J Urol. 2004 Aug;172(2):533-6. doi: 10.1097/01.ju.0000132388.54703.4d. PMID 15247722
- [Background] Sant GR, Propert KJ, Hanno PM, Burks D, Culkin D, Diokno AC, Hardy C, Landis JR, Mayer R, Madigan R, Messing EM, Peters K, Theoharides TC, Warren J, Wein AJ, Steers W, Kusek JW, Nyberg LM; Interstitial Cystitis Clinical Trials Group. A pilot clinical trial of oral pentosan polysulfate and oral hydroxyzine in patients with interstitial cystitis. J Urol. 2003 Sep;170(3):810-5. doi: 10.1097/01.ju.0000083020.06212.3d. PMID 12913705
- [Background] Lee B, Elston DM. The uses of naltrexone in dermatologic conditions. J Am Acad Dermatol. 2019 Jun;80(6):1746-1752. doi: 10.1016/j.jaad.2018.12.031. Epub 2018 Dec 21. PMID 30582992
- [Background] Tortelly VD, De Mattos T, Fernandes LSA, Nunes BEM, Melo DF. Low-dose naltrexone: a novel adjunctive treatment in symptomatic alopecias? Dermatol Online J. 2019 Aug 15;25(8):13030/qt6j45h81f. PMID 31553867
- [Background] Zashin S. Sjogren's Syndrome: Clinical Benefits of Low-dose Naltrexone Therapy. Cureus. 2019 Mar 11;11(3):e4225. doi: 10.7759/cureus.4225. PMID 31123647
- [Background] Trofimovitch D, Baumrucker SJ. Pharmacology Update: Low-Dose Naltrexone as a Possible Nonopioid Modality for Some Chronic, Nonmalignant Pain Syndromes. Am J Hosp Palliat Care. 2019 Oct;36(10):907-912. doi: 10.1177/1049909119838974. Epub 2019 Mar 27. PMID 30917675
- [Background] Jaros J, Lio P. Low Dose Naltrexone in Dermatology. J Drugs Dermatol. 2019 Mar 1;18(3):235-238. PMID 30909326
- [Background] Cui X, Jing X, Lutgendorf SK, Bradley CS, Schrepf A, Erickson BA, Magnotta VA, Ness TJ, Kreder KJ, O'Donnell MA, Luo Y. Cystitis-induced bladder pain is Toll-like receptor 4 dependent in a transgenic autoimmune cystitis murine model: a MAPP Research Network animal study. Am J Physiol Renal Physiol. 2019 Jul 1;317(1):F90-F98. doi: 10.1152/ajprenal.00017.2019. Epub 2019 May 15. PMID 31091120
- [Background] Suskind AM, Berry SH, Suttorp MJ, Elliott MN, Hays RD, Ewing BA, Clemens JQ. Health-related quality of life in patients with interstitial cystitis/bladder pain syndrome and frequently associated comorbidities. Qual Life Res. 2013 Sep;22(7):1537-41. doi: 10.1007/s11136-012-0285-5. Epub 2012 Oct 7. PMID 23054497
- [Background] Toljan K, Vrooman B. Low-Dose Naltrexone (LDN)-Review of Therapeutic Utilization. Med Sci (Basel). 2018 Sep 21;6(4):82. doi: 10.3390/medsci6040082. PMID 30248938
- [Background] Oaks Z, Stage A, Middleton B, Faraone S, Johnson B. Clinical utility of the cold pressor test: evaluation of pain patients, treatment of opioid-induced hyperalgesia and fibromyalgia with low dose naltrexone. Discov Med. 2018 Nov;26(144):197-206. PMID 30695679
- [Background] Patten DK, Schultz BG, Berlau DJ. The Safety and Efficacy of Low-Dose Naltrexone in the Management of Chronic Pain and Inflammation in Multiple Sclerosis, Fibromyalgia, Crohn's Disease, and Other Chronic Pain Disorders. Pharmacotherapy. 2018 Mar;38(3):382-389. doi: 10.1002/phar.2086. Epub 2018 Feb 23. PMID 29377216
- [Background] Parkitny L, Younger J. Reduced Pro-Inflammatory Cytokines after Eight Weeks of Low-Dose Naltrexone for Fibromyalgia. Biomedicines. 2017 Apr 18;5(2):16. doi: 10.3390/biomedicines5020016. PMID 28536359
- [Background] Hota D, Srinivasan A, Dutta P, Bhansali A, Chakrabarti A. Off-Label, Low-Dose Naltrexone for Refractory Painful Diabetic Neuropathy. Pain Med. 2016 Apr;17(4):790-1. doi: 10.1093/pm/pnv009. Epub 2015 Dec 7. No abstract available. PMID 26814245
- [Background] Younger J, Noor N, McCue R, Mackey S. Low-dose naltrexone for the treatment of fibromyalgia: findings of a small, randomized, double-blind, placebo-controlled, counterbalanced, crossover trial assessing daily pain levels. Arthritis Rheum. 2013 Feb;65(2):529-38. doi: 10.1002/art.37734. PMID 23359310
- [Background] Ramanathan S, Panksepp J, Johnson B. Is fibromyalgia an endocrine/endorphin deficit disorder? Is low dose naltrexone a new treatment option? Psychosomatics. 2012 Nov-Dec;53(6):591-4. doi: 10.1016/j.psym.2011.11.006. Epub 2012 Apr 4. No abstract available. PMID 22480625
- [Background] de Oliveira MG, Monica FZ, Calmasini FB, Alexandre EC, Tavares EBG, Soares AG, Costa SKP, Antunes E. Deletion or pharmacological blockade of TLR4 confers protection against cyclophosphamide-induced mouse cystitis. Am J Physiol Renal Physiol. 2018 Sep 1;315(3):F460-F468. doi: 10.1152/ajprenal.00100.2018. Epub 2018 May 2. PMID 29717937
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Ghai B, Bansal D, Hota D, Shah CS. Off-label, low-dose naltrexone for refractory chronic low back pain. Pain Med. 2014 May;15(5):883-4. doi: 10.1111/pme.12345. No abstract available. PMID 24967470
- [Background] Younger J, Parkitny L, McLain D. The use of low-dose naltrexone (LDN) as a novel anti-inflammatory treatment for chronic pain. Clin Rheumatol. 2014 Apr;33(4):451-9. doi: 10.1007/s10067-014-2517-2. Epub 2014 Feb 15. PMID 24526250
- [Background] Chopra P, Cooper MS. Treatment of Complex Regional Pain Syndrome (CRPS) using low dose naltrexone (LDN). J Neuroimmune Pharmacol. 2013 Jun;8(3):470-6. doi: 10.1007/s11481-013-9451-y. Epub 2013 Apr 2. PMID 23546884
- [Background] Frech T, Novak K, Revelo MP, Murtaugh M, Markewitz B, Hatton N, Scholand MB, Frech E, Markewitz D, Sawitzke AD. Low-dose naltrexone for pruritus in systemic sclerosis. Int J Rheumatol. 2011;2011:804296. doi: 10.1155/2011/804296. Epub 2011 Sep 12. PMID 21918649
- [Background] Cree BA, Kornyeyeva E, Goodin DS. Pilot trial of low-dose naltrexone and quality of life in multiple sclerosis. Ann Neurol. 2010 Aug;68(2):145-50. doi: 10.1002/ana.22006. PMID 20695007
- [Background] Sharafaddinzadeh N, Moghtaderi A, Kashipazha D, Majdinasab N, Shalbafan B. The effect of low-dose naltrexone on quality of life of patients with multiple sclerosis: a randomized placebo-controlled trial. Mult Scler. 2010 Aug;16(8):964-9. doi: 10.1177/1352458510366857. Epub 2010 Jun 9. PMID 20534644
- [Background] Younger J, Mackey S. Fibromyalgia symptoms are reduced by low-dose naltrexone: a pilot study. Pain Med. 2009 May-Jun;10(4):663-72. doi: 10.1111/j.1526-4637.2009.00613.x. Epub 2009 Apr 22. PMID 19453963
- [Background] Gironi M, Martinelli-Boneschi F, Sacerdote P, Solaro C, Zaffaroni M, Cavarretta R, Moiola L, Bucello S, Radaelli M, Pilato V, Rodegher M, Cursi M, Franchi S, Martinelli V, Nemni R, Comi G, Martino G. A pilot trial of low-dose naltrexone in primary progressive multiple sclerosis. Mult Scler. 2008 Sep;14(8):1076-83. doi: 10.1177/1352458508095828. PMID 18728058
- [Background] Kariv R, Tiomny E, Grenshpon R, Dekel R, Waisman G, Ringel Y, Halpern Z. Low-dose naltreoxone for the treatment of irritable bowel syndrome: a pilot study. Dig Dis Sci. 2006 Dec;51(12):2128-33. doi: 10.1007/s10620-006-9289-8. Epub 2006 Nov 1. PMID 17080248
- [Background] Majumdar SR, Roe MT, Peterson ED, Chen AY, Gibler WB, Armstrong PW. Better outcomes for patients treated at hospitals that participate in clinical trials. Arch Intern Med. 2008 Mar 24;168(6):657-62. doi: 10.1001/archinternmed.2007.124. PMID 18362259
- [Background] Meske DS, Lawal OD, Elder H, Langberg V, Paillard F, Katz N. Efficacy of opioids versus placebo in chronic pain: a systematic review and meta-analysis of enriched enrollment randomized withdrawal trials. J Pain Res. 2018 May 3;11:923-934. doi: 10.2147/JPR.S160255. eCollection 2018. PMID 29765246
- [Background] Hale M, Khan A, Kutch M, Li S. Once-daily OROS hydromorphone ER compared with placebo in opioid-tolerant patients with chronic low back pain. Curr Med Res Opin. 2010 Jun;26(6):1505-18. doi: 10.1185/03007995.2010.484723. PMID 20429852
- [Background] Schwartz S, Etropolski M, Shapiro DY, Okamoto A, Lange R, Haeussler J, Rauschkolb C. Safety and efficacy of tapentadol ER in patients with painful diabetic peripheral neuropathy: results of a randomized-withdrawal, placebo-controlled trial. Curr Med Res Opin. 2011 Jan;27(1):151-62. doi: 10.1185/03007995.2010.537589. PMID 21162697
- See also: Amitriptyline: Drug information. Accessed 10/29/2019 — https://www-uptodate-com.proxy.uchicago.edu/contents/amitriptyline-drug-
- See also: Management of interstitial cystitis/bladder pain syndrome. Uptpdate. Accessed 12/5/2019 — https://www-uptodate-com.proxy.uchicago.edu/contents/management-of-interstitial-cystitis-bladder-pain-syndrome?source=history_widget#H285129

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low-dose Naltrexone | Placebo
Started | 1 | 2
Completed | 1 | 1
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-dose Naltrexone | Placebo | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 | 52 (8.5) | 52 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Interstitial Cystitis Symptom Index
Description: The effect of LDN (low-dose naltrexone) in decreasing symptoms associated with IC/PBS (interstitial cystitis/painful bladder syndrome) when treating with low-dose naltrexone as scored by the Interstitial Cystitis Symptom Index as compared to placebo. Scores are from 0 to 20, with lower scores indicating less symptoms associated with IC/PBS.
Time Frame: six weeks
Population: Excluding one participant who withdrew from the study.
Measure: Number; unit: score on a scale
Arm/Group | Low-dose Naltrexone | Placebo
Number analyzed (Participants) | 1 | 1
score on a scale | 6 | 5

2. Primary Outcome: Visual Analog Scale
Description: The effect of LDN in decreasing pain associated with IC/PBS when treating with low-dose naltrexone as scored by visual analog scale as compared with placebo. Scores are from 0 to 10, with lower scores indicating less pain.
Time Frame: six weeks
Population: Excluding one participant who withdrew from the study.
Measure: Number; unit: score on a scale
Arm/Group | Low-dose Naltrexone | Placebo
Number analyzed (Participants) | 1 | 1
score on a scale | 0 | 0

3. Secondary Outcome: Change in Interstitial Cystitis Problem Index
Description: The changes in IC/PBS associated problems when treating interstitial cystitis/painful bladder syndrome with low-dose naltrexone as scored by the Interstitial Cystitis Problem Index, prior to initiating treatment and at the conclusion of 6 weeks of treatment. Scores are from 0-16, with lower scores indicating a better score, with fewer problems associated with IC/PBS. The change was calculated from two time points as the value prior to initiating treatment minus the value at the conclusion of 6 weeks of treatment.
Time Frame: prior to initiating treatment and at the conclusion of 6 weeks of treatment
Population: Excluding one participant who withdrew from the study.
Measure: Number; unit: score on a scale
Arm/Group | Low-dose Naltrexone | Placebo
Number analyzed (Participants) | 1 | 1
score on a scale | 4 | 11

4. Secondary Outcome: Change in Urinary Frequency
Description: The change in number of patient voids during the day when comparing LDN against placebo as determined from 24 hour bladder diary performed by patient prior to initiating treatment and at the conclusion of 6 weeks of treatment. The change was calculated from two time points as the value prior to initiating treatment minus the value at the conclusion of 6 weeks of treatment.
Time Frame: prior to initiating treatment and at the conclusion of 6 weeks of treatment
Population: Excluding one participant who withdrew from the study.
Measure: Number; unit: voids per day
Arm/Group | Low-dose Naltrexone | Placebo
Number analyzed (Participants) | 1 | 1
voids per day | 8 | 11

5. Secondary Outcome: Change in Number of Nocturia
Description: The change in number of patient voids during at night when comparing LDN against placebo as determined from 24 hour bladder diary performed by patient prior to initiating treatment and at the conclusion of 6 weeks of treatment. The change was calculated from two time points as the value prior to initiating treatment minus the value at the conclusion of 6 weeks of treatment.
Time Frame: prior to initiating treatment and at the conclusion of 6 weeks of treatment
Population: Excluding one participant who withdrew from the study.
Measure: Number; unit: voids per night
Arm/Group | Low-dose Naltrexone | Placebo
Number analyzed (Participants) | 1 | 1
voids per night | 3 | 2

6. Secondary Outcome: Change in Pelvic Pain and Urgency/Frequency Symptoms
Description: The change in pelvic pain and urgency/frequency symptoms as measured on the Pelvic Pain and Urgency/Frequency Patient Symptom Scale, prior to initiating treatment and at the conclusion of 6 weeks of treatment. Scores can range from 0-23, with higher scores indicating more severe symptoms associated with IC/PBS. The change was calculated from two time points as the value prior to initiating treatment minus the value at the conclusion of 6 weeks of treatment.
Time Frame: prior to initiating treatment and at the conclusion of 6 weeks of treatment
Population: Excluding one participant who withdrew from the study.
Measure: Number; unit: score on a scale
Arm/Group | Low-dose Naltrexone | Placebo
Number analyzed (Participants) | 1 | 1
score on a scale | 3 | 7

7. Secondary Outcome: Change in Pelvic Pain and Urgency/Frequency Bother
Description: The change in pelvic pain and urgency/frequency bother as measured on the Pelvic Pain and Urgency/Frequency Patient Symptom Scale, prior to initiating treatment and at the conclusion of 6 weeks of treatment. Scores can range from 0-12, with higher values corresponding to more bother from IC/PBS symptoms. The change was calculated from two time points as the value prior to initiating treatment minus the value at the conclusion of 6 weeks of treatment.
Time Frame: prior to initiating treatment and at the conclusion of 6 weeks of treatment
Population: Excluding one participant who withdrew from the study.
Measure: Number; unit: score on a scale
Arm/Group | Low-dose Naltrexone | Placebo
Number analyzed (Participants) | 1 | 1
score on a scale | 1 | 7

8. Secondary Outcome: Patient Perceived Quality of Life: SF-36
Description: Patient perceived quality of life as measured by the medical outcomes study short form 36 (SF-36). Higher scores indicate a more favorable health status. There are 8 subscales, which when averaged, include a score from 0-100.
Time Frame: six weeks
Population: Excluding one participant who withdrew from the study.
Measure: Number; unit: score on a scale
Arm/Group | Low-dose Naltrexone | Placebo
Number analyzed (Participants) | 1 | 1
score on a scale | 86 | 84

9. Secondary Outcome: Adverse Effects
Description: The percentage of patients complaining of adverse effects from LDN including vivid dreams, nightmares, insomnia, GI disturbances such as stomach cramps or diarrhea, agitation, anxiety, flu-like symptoms and headaches.
Time Frame: six weeks
Population: Excluding one participant who withdrew from the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-dose Naltrexone | Placebo
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

10. Secondary Outcome: Medication Tolerability
Description: The percentage of patients who discontinue the study medication measured by the tolerability survey.
Time Frame: six weeks
Population: Excluding one participant who withdrew from the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-dose Naltrexone | Placebo
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

11. Secondary Outcome: Number of Days With Pain Medications
Description: The number of days with pain medication use while using LDN, as determined by a pain medication diary.
Time Frame: six weeks
Population: Excluding one participant who withdrew from the study.
Measure: Number; unit: days
Arm/Group | Low-dose Naltrexone | Placebo
Number analyzed (Participants) | 1 | 1
days | 13 | 42

ADVERSE EVENTS:
Time Frame: At two weeks and at four weeks, an average up to six weeks
Description: No adverse event was recorded for the three participants enrolled in the study.
Arm/Group | Low-dose Naltrexone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-18): https://cdn.clinicaltrials.gov/large-docs/72/NCT04313972/Prot_SAP_000.pdf